CLINICAL TRIAL: NCT06350344
Title: Smart Technology Facilitated Patient-centered Venous Thromboembolism Management: A Multicenter Cohort Study
Brief Title: Smart Technology Facilitated Patient-centered Venous Thromboembolism Management
Acronym: SmaVTE-COR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HZKY-PJ-2024-8-2
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-03

CONDITIONS: Venous Thromboembolism; Digital Health; Health Education
Keywords: Venous Thromboembolism; Mobile Health; Prophylaxis; Health Education
MeSH Terms: conditions — Venous Thromboembolism; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mVTEA Management Group (Experimental): Patients with high-risk of VTE will be discharged with mVTEA-assisted patient-centered VTE management.
  Interventions: Device: mobile venous thromboembolism application (mVTEA)

INTERVENTIONS:
Device: mobile venous thromboembolism application (mVTEA) — mVTEA will assist in the management of patients with high-risk of VTE during the post-hospitalization follow-up phase. The mVTEA's doctor terminal automatically sends VTE-related health education materials in different frequencies and contents based on the patient's knowledge of VTE prevention and treatment, as well as their risk of thrombosis and bleeding during follow-up. In addition, thrombosis physicians on the mVTEA's doctor terminal can deliver health education to patients based on their condition. This can be done through the mVTEA doctor-patient communication module, which includes text, voice, and video communication.

SUMMARY:
Smart technologies, such as wearable devices, mobile technologies, and artificial intelligence, are being investigated for use in health management. These technologies have the potential to be applied in disease pre-warning, decision-making support, health education, and healthcare maintenance. They are expected to address the challenges in managing thrombosis, improve access to high-quality medical resources in various regions, and enhance the development of a network for thrombosis rescue and treatment prevention.

The objective of this study is to observe the long-term effect of mobile venous thromboembolism application (mVTEA) based patient-centered management of venous thromboembolism (VTE) on thromboprophylaxis, and establish a foundation of evidence for managing patients with high-risk VTE.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients ≥18 years of age at admission;
* At high-risk of VTE at discharge: Padua score ≥4 for medical patients and Caprini score ≥5 for surgical patients;
* Signed informed consent.

Exclusion Criteria:

* Diagnosis of VTE at discharge;
* Mental disorder or combination of other serious diseases leading to incapacity for independent living;
* Inability to use smartphones, computer tablets and other smart devices;
* Being pregnant or breastfeeding;
* Have participated in similar trials or are undergoing other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2353 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
VTE-related composite event | At 1-year follow-up
  The primary outcome was the occurrence of VTE-related composite event at 1-year follow-up, which was defined as a composite of VTE, major bleeding, VTE-related hospitalization, and all-cause death.

SECONDARY OUTCOMES:
VTE-KAP questionnaire score | At 3, 12, and 24-month follow-up
  The VTE-KAP questionnaire is a self-administered questionnaire that includes demographic characteristics, knowledge, attitude, and practice (KAP) of patients towards VTE prevention and treatment. The VTE-KAP questionnaire consists of a total of 53 questions with an overall score range of 41 to 283. The higher the score, the higher the level of knowledge, attitude, and practice. The VTE-KAP questionnaire scores of the patients regarding the prevention and treatment of VTE will be evaluated at 3, 12, and 24-month follow-up.
Generic quality of life | At 3, 12, and 24-month follow-up
  Generic, non-disease-speciﬁc health-related quality of life (QoL) is assessed using the EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire and its corresponding visual analogue scale at 3, 12, and 24-month follow-up. Brieﬂy, the EQ-5D-5L generates an overall index that ranges from 0 (lowest generic QoL) to 1 (highest generic QoL) and is calculated based on country-speciﬁc reference value sets. The EQ-5D-5L health index was calculated with the value set for China. The EuroQol visual analogue scale ranges from 0 to 100, with higher scores indicating better health.
VTE events | At 3, 6, 12, and 24-month follow-up
  VTE events will be documented during the follow-up. VTE events are categorized into two groups: new-onset VTE, and hospital-acquired VTE (HA-VTE).
  VTE that occurred for the first time during the study period, including deep vein thrombosis (DVT) and pulmonary embolism (PE), is classified as new-onset VTE.
  HA-VTE is defined as any new-onset VTE that has occurred within 90 days of hospital discharge.
Major bleeding | At 3, 6, 12, and 24-month follow-up
  The major bleeding events as defined by the International Society on Thrombosis and Hemostasis (ISTH) will be documented during the follow-up.
VTE-related hospitalization | At 3, 6, 12, and 24-month follow-up
  Hospitalization due to the new-onset DVT and/or PE will be documented during the follow-up.
New-onset of atrial fibrillation or atrial flutter | At 3, 6, 12, and 24-month follow-up
  The new-onset of atrial fibrillation or atrial flutter will be documented during the follow-up.
Death | At 3, 6, 12, and 24-month follow-up
  Death will be documented during the follow-up. It is categorized into all-cause death and PE-related death. All-cause death is defined as death that occurs during the study period, regardless of cause.PE-related death is defined as death that is unequivocally due to PE.

CONTACTS AND LOCATIONS:
Overall Officials: YU-TAO GUO, Doctor, Study Chair — Sixth Medical Center of Chinese PLA General Hospital
Locations (1):
- Sixth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chew HK, Davies AM, Wun T, Harvey D, Zhou H, White RH. The incidence of venous thromboembolism among patients with primary lung cancer. J Thromb Haemost. 2008 Apr;6(4):601-8. doi: 10.1111/j.1538-7836.2008.02908.x. Epub 2008 Jan 17. PMID 18208538
- [Background] Kang MJ, Ryoo BY, Ryu MH, Koo DH, Chang HM, Lee JL, Kim TW, Kang YK. Venous thromboembolism (VTE) in patients with advanced gastric cancer: an Asian experience. Eur J Cancer. 2012 Mar;48(4):492-500. doi: 10.1016/j.ejca.2011.11.016. Epub 2011 Dec 12. PMID 22169121
- [Background] Henke PK, Kahn SR, Pannucci CJ, Secemksy EA, Evans NS, Khorana AA, Creager MA, Pradhan AD; American Heart Association Advocacy Coordinating Committee. Call to Action to Prevent Venous Thromboembolism in Hospitalized Patients: A Policy Statement From the American Heart Association. Circulation. 2020 Jun 16;141(24):e914-e931. doi: 10.1161/CIR.0000000000000769. Epub 2020 May 7. PMID 32375490